CLINICAL TRIAL: NCT00043199
Title: A Phase II Study of Aroplatin in Subjects With Recurrent, Unresectable and Metastatic Colorectal Cancer Refractory to 5-Fluorouracil (5-FU)/Leucovorin or Capecitabine, and Irinotecan
Brief Title: A Safety and Effectiveness Study of Aroplatin in Patients With Advanced Colorectal Cancer Resistant to Standard Therapies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aronex Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-726-01
Record Dates: First submitted 2002-08-06; First posted 2002-08-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumor; Neoplasms, Colorectal; Unresectable; Metastatic; Refractory
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II)

INTERVENTIONS:
Drug: Aroplatin (Liposomal NDDP, L-NDDP)

SUMMARY:
To determine the rate of response and duration of reponse following therapy with Aroplatin in subjects with advanced colorectal cancer resistant to standard therapies. Secondary objectives are to determine safety and tolerability of the Aroplatin therapy.

DETAILED DESCRIPTION:
Primary Objective:

* To determine response rate (RR; complete and partial response[CR,PR] and duration after therapy with Aroplatin (Liposomal NDDP, L-NDDP) in subjects with locally recurrent, unresectable or metastatic colorectal cancer refractory to 5-FU/leucovorin or capecitabine, and irinotecan.

Secondary Objective:

* To determine safety and tolerability of the Aroplatin therapy.

This is a single-arm, open-label phase II study. Subjects refractory to 5-FU/leucovorin or capecitabine, and irinotecan therapies will be enrolled. Dosing will be every four weeks with individual dose escalations and adjustments for toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer, locally recurrent, unresectable or metastatic disease (AJCC);
* Measurable disease (RECIST criteria);
* Cancer refractory to 5-FU/leucovorin or capecitabine, and irinotecan;
* ECOG performance score of 0-2;
* Adequate hematopoietic, liver and renal function;
* Adequate cardiac function (maximum of class II, NYHA);
* Women of child-bearing potential must have a negative urine or serum pregnancy test;
* Signed written informed consent;
* Subjects must be willing to to be followed during the course of treatment/observation and follow-up.

Exclusion Criteria:

* Other malignancies treated within the last five years, except in situ cervix carcinoma or non-melanoma skin cancer;
* Pregnant or breast feeding subjects, or male or female subjects of child producing potential who will not agree to use adequate contraception during the treatment phase of the study;
* Prior therapy with oxaliplatin;
* Known brain metastases;
* Active, uncontrolled infection or other serious medical illnesses;
* Subjects may not be using or have used any investigational therapy during four weeks before start of the protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Cancer Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona